CLINICAL TRIAL: NCT02695550
Title: Study of Safety, Efficacy and Pharmacokinetics of CT-707 in Patients With ALK-positive Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centaurus Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-707-101
Record Dates: First submitted 2016-02-23; First posted 2016-03-01 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — conteltinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CT-707 (Experimental): ALK-positive non-small cell lung cancer resistant to Crizotinib treatment
  Interventions: Drug: CT-707

INTERVENTIONS:
Drug: CT-707

SUMMARY:
This is a Phase I study of the ALK/FAK/Pyk2 inhibitor CT-707 in patients with ALK-positive non-small cell lung cancer.

The purpose of the study is to determine the MTD/RP2D of CT-707 and evaluate whether CT-707 is safe and has beneficial effects in ALK-positive advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients must be diagnosed with ALK-positive advanced NSCLC. The tumor must be ALK-positive as determined by ALK rearrangement in ≥15% of cells (as measured by FISH using the Vysis break-apart ALK probe) or by using the Ventana ALK IHC test. The analysis may be performed locally.

Eastern cooperative oncology group (ECOG) performance status ≤ 2. Measurable disease as per RECIST v1.1

Availability of tumor sample:

Exclusion Criteria:

Patients with symptomatic central nervous system (CNS) metastases who are neurologically unstable or require increasing doses of steroids or local CNS-directed therapy to control their CNS disease Impaired cardiac function or any clinically significant cardiac disease Patients with abnormal laboratory values during screening and on day 1 of pre-dose Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of CT-707 Patient has a history of pancreatitis or history of increased amylase or lipase that was due to pancreatic disease.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of dose limiting toxicities (DLTs) during the first cycle of treatment (Phase I) | 28 days
  Maximum Tolerated Dose(s) (MTD(s)) and/or recommended phase 2 dose (RP2D(s)) of CT-707 in ALK-positive non-small cell lung cancer (NSCLC) patients. Cycle = 28 days
Frequency of adverse events/serious adverse events | Up to 24 months
  Characterization of the safety and tolerability of CT-707 as determined by changes in laboratory values and electrocardiograms

SECONDARY OUTCOMES:
Overall Response Rate (ORR) - Phase I | Up to 24 month
  Preliminary measure of anti-tumor activity of CT-707
Progression free survival (PFS) per RECIST v1.1 - Phase I | Up to 24 months
  Preliminary measures of anti-tumor activity of CT-707
Duration of response (DOR) | Up to 24 months
  Preliminary measure of anti-tumor activity of CT-707

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Dr, Principal Investigator — Cancer Hospital of Chines Academy of Medical Sciences
Locations (1):
- Cancer Hospital of Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xing P, Zhao Q, Zhang L, Wang H, Huang D, Hu P, Sun Y, Shi Y. Conteltinib (CT-707) in patients with advanced ALK-positive non-small cell lung cancer: a multicenter, open-label, first-in-human phase 1 study. BMC Med. 2022 Nov 23;20(1):453. doi: 10.1186/s12916-022-02646-0. PMID 36424628
- [Derived] Liang C, Zhang N, Tan Q, Liu S, Luo R, Wang Y, Shi Y, Han X. CT-707 Overcomes Resistance of Crizotinib through Activating PDPK1- AKT1 Pathway by Targeting FAK. Curr Cancer Drug Targets. 2019;19(8):655-665. doi: 10.2174/1568009618666181031152140. PMID 30381078